CLINICAL TRIAL: NCT00382434
Title: The ED Pharmacist as a Safety Measure in Emergency Medicine
Brief Title: Emergency Pharmacist Safety Study
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Other Study IDs: 1U18HS015818 (AHRQ); RSRB #11834
Record Dates: First submitted 2006-09-27; First posted 2006-09-29 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Adverse Drug Event, Potential Adverse Drug Event, and Quality Measures
Keywords: emergency pharmacist; emergency medicine; emergency department; medical error; adverse event; pharmacist; patient safety
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Emergencies

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EPh Present: the emergency pharmacist is present in the ED when the medical care is provided
  Interventions: Procedure: presence of an emergency pharmacist in the ED

INTERVENTIONS:
Procedure: presence of an emergency pharmacist in the ED

SUMMARY:
The Emergency Department (ED) is a unique environment in medicine, and many safety mechanisms used in other hospital settings cannot be applied in the ED. For example, clinical pharmacists have traditionally provided extra layers of protection to hospital inpatients by cross-checking provider orders for appropriate dosing, contraindications, and interactions. Because medications in the ED must be accessed immediately and are often one-time doses, the use of central pharmacy services would introduce an unacceptable delay to the administration of medication. Although some hospitals have programs in place in which a pharmacist responds to the ED for cardiac arrests or trauma team activations, few have reported programs which involve a clinical pharmacist assigned exclusively to the emergency department. Nonetheless, published reports have asserted that ED-based pharmacists can increase patient safety. Although this concept appears logical, no study has attempted to show that these programs reduce potential adverse drug events in the ED. We propose to implement and optimize an ED Pharmacist (EDP) program as a safe practice intervention in a large ED. The hospital has provided funding for two permanent full time positions starting at the beginning of the award period. In the initial phase interviews of physicians, nurses, pharmacists, and patients will be conducted and the results will be used to optimize the EDP role. A large-scale chart review study will then be conducted to evaluate whether there is a reduction in frequency of potential and adverse drug events during times that the EDP is on duty. Staff perceptions of the effectiveness of this program will also be evaluated. The overall goal of this initiative is to create an effective EDP program that will decrease the rate of adverse drug events in ED patients, and to create a "toolkit" to facilitate the introduction of similar programs into other EDs. This toolkit will include a description of the formal, optimized role of the EDP, challenges and solutions in implementation, and evidence to support the efficacy of such a program.

ELIGIBILITY:
Inclusion Criteria:

* pediatric (less than 19), geriatric (>64), or critically ill (all ages)

Exclusion Criteria:

* investigator involved or incomplete chart

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: emergency department patients
Sampling Method: Probability Sample
Enrollment: 10224 (Actual)
Dates: Start 2005-08; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rollin J Fairbanks, MD, MS, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States